CLINICAL TRIAL: NCT02902562
Title: Quantitative Assessment of Synovitis and Therapy Response in Inflammatory Arthritis With Contrast Enhanced Ultrasound
Brief Title: Synovitis and Therapy Response in Inflammatory Arthritis With Contrast Enhanced Ultrasound
Acronym: CEUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Wright Foundation (Unknown)
Responsible Party: Principal Investigator, George Matcuk, Associate Professor, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HS-15-00377
Record Dates: First submitted 2016-08-29; First posted 2016-09-16 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Synovitis; Rheumatoid Arthritis
MeSH Terms: conditions — Synovitis; Arthritis, Rheumatoid | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study Visit (Other): You will have a Contrast Enhanced Ultrasound (CEUS) and contrast Magnetic Resonance Imaging (MRI) which will take about 2 hours.
  Interventions: Procedure: Contrast Enhanced Ultrasound (CEUS); Procedure: Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Procedure: Contrast Enhanced Ultrasound (CEUS) — An intravenous line (IV) line will be inserted into a vein in your arm. You will be asked to lie on a table for the ultrasound imaging. First, a regular ultrasound (without contrast) will be performed and the images will be recorded. For the contrast enhanced ultrasound, the contrast agent will be injected into your IV line. We will perform another ultrasound and the images will be recorded
Procedure: Magnetic Resonance Imaging (MRI) — For the contrast MRI, the contrast agent will be injected into your IV line The MRI scanner is a small, tunnel-like machine in which a patient will be required to lie still for a long period of time. There is little space inside the scanner, which causes anxiety and discomfort for patients who fear enclosed spaces. A technician will be present at all times during the examination to communicate with you about how you are feeling.

SUMMARY:
This study is about using contrast-enhanced ultrasound (CEUS) to assess the degree of synovitis (joint inflammation) in patients with inflammatory arthritis, such as rheumatoid arthritis, and whether it can be used for assessing a treatment response. The investigators hope to learn whether contrast enhanced ultrasounds are better than regular imaging techniques, such as MRI, when used to evaluate the response to disease modifying anti-rheumatic drug (DMARD) therapy in inflammatory arthritis.

DETAILED DESCRIPTION:
Inflammatory arthritis affects approximately 1% of the world population and can lead to significant pain and disability. Although radiographs can identify characteristic patterns of joint space narrowing and erosive changes, these findings are typically late findings and represent irreversible damage. With the development of disease modifying anti-rheumatic drugs (DMARDs), the goal is now to identify the pre-erosive inflammatory features and identify the patients that progress further into severe functional debility if not treated immediately.

MRI with gadolinium enhancement is proven to be very effective in early detection of soft tissue, bone erosions, synovitis, the integrity of ligaments, cartilage and bone marrow edema. However, MRI is expensive, may be impractical for assessing multiple joints and has relatively long examination time. Some patients may have claustrophobia and some may have contraindications to gadolinium administration. The investigators overarching goal is to determine whether the perfusion information provided by novel ultrasound based techniques such as, contrast enhanced ultrasound and superb microvascular imaging, can be used for assessment of treatment response to DMARD therapy for inflammatory arthritis. The recent advances in evaluation of vascularity of the tumors using contrast ultrasound technique can also be applied to rheumatological diseases. It is ideal to develop a sensitive imaging technique that can be routinely available and is relatively cheap. Ultrasound is available and has low cost and can be used for assessment of treatment response to DMARD therapy

ELIGIBILITY:
Inclusion Criteria:

* Patients (≥ 18 years of age) that meet diagnostic criteria for an inflammatory arthritis.
* Clinical suspicion of active synovitis involving at least one target joint.
* Patients competent to sign study specific Informed Consent.
* Patients willing to comply with protocol requirements.
* Intent to treat with disease-modifying anti-rheumatic drugs (DMARDs).

Exclusion Criteria:

* Patients who are pregnant or less than 18 years of age.
* Patients who have a known cardiac shunt or pulmonary hypertension.
* Patients with any known hypersensitivity to perflutren or gadolinium contrast agents or renal insufficiency (GFR < 30 mL/min).
* Patients who cannot consent for themselves.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-08-31 (Actual); Primary Completion 2018-07-17 (Actual); Study Completion 2018-08-22 (Actual)

PRIMARY OUTCOMES:
Kappa coefficient | 12 months
  To assess the inter-reader agreement as well as the agreement between CEUS versus MRI determined treatment response.

CONTACTS AND LOCATIONS:
Overall Officials: George R Matcuk, MD, Principal Investigator — University of Southern California
Locations (1):
- USC Department of Radiology, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided